CLINICAL TRIAL: NCT04869436
Title: The 'Real World' Olfactory Outcomes Treating Nasal Polyposis With Dupilumab
Brief Title: Olfactory Outcomes of Dupilumab Treatment for Nasal Polyposis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Leigh Sowerby, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3618
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Olfactory Disorder
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Single group 6 months treatment with Dupilumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dupilumab group (Experimental): Patients with CRSwNP will have an initial dose of 600 mg of dupilumab, and 5 additional doses of 300mg every 4 weeks for 6 months.
  Interventions: Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT]

INTERVENTIONS:
Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT] — Dupilumab will be administered subcutaneously for 6 months (1 initial 600mg dose + 5 300mg doses every 4 weeks)

SUMMARY:
The study aims to investigate the olfactory TDI score (Threshold, Discrimination, Identification) using the Sniffin' sticks test for patients with chronic rhinosinusitis with nasal polyps (CRSwNP) on dupilumab. Twenty-seven adult patients will be followed up during the treatment with dupilumab on three visits to the Otolaryngology Clinic (Baseline, 3 months and 6 months).

The primary endpoint will be the TDI score. Nasal polyp score, Quality of Olfactory Disorders - negative symptoms (QOD-NS symptom scores), SNOT-22 will be secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Chronic rhinosinusitis with Nasal Polyps
* Olfactory loss
* Clinical indication for treatment with Dupilumab

Exclusion Criteria:

Patients with olfactory loss from other causes such as:

* Sinonasal malignancies
* Trauma
* Idiopathic olfactory loss
* Use of cocaine
* COVID-19 related olfactory loss
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Smell Threshold, Identification and Discrimination (TDI score) at week 12 and week 24. | Baseline, 12 weeks and 24 weeks.
  The Sniffin' Sticks test involves testing odor for threshold and discrimination whilst blind folded and secondly odor identification. The sum of four odors responses ranges from 0-16. The sum of total score from odor Threshold, Discrimination and Identification (TDI) is a maximum of 48 points. The total score is graded as; normosmia equals or over 30.5 points, hyposmia 16.5-30 points and anosmia less than 16.5 points.

SECONDARY OUTCOMES:
Change from Baseline in the Nasal Polyps score at weeks 12 and 24. | Baseline, 12 weeks and 24 weeks.
  Nasal Polyps score is the sum of the right and left nostril scores (endoscopic assessment). Total score ranges from 0 (no polyps) to 8 (large polyps on for each nostril [4+4] ).
Change from Baseline in the Sino-nasal outcome test- 22 (SNOT-22) at weeks 12 and 24. | Baseline, 12 weeks and 24 weeks.
  SNOT-22 is a validated questionnaire to assess the impact of chronic rhinosinusitis on patients' quality of life. Patient grades the impact of 22 potential symptoms in their life, by choosing from 0 [no problem] to 5 [problem as bad as it can be]. Highest possible score is 10 (worst quality of life); minimal clinically important change ≥ 8.90
Change from Baseline in the QOD-NS at weeks 12 and 24. | Baseline, 12 weeks and 24 weeks.
  Quality of Olfactory Disorders - negative symptoms (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh J Sowerby, MD, FRCS, Principal Investigator — St. Joseph's Hospital London, ON, Canada
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available.